CLINICAL TRIAL: NCT02827708
Title: Efficacy and Safety of Oral Semaglutide Versus Placebo in Subjects With Type 2 Diabetes and Moderate Renal Impairment
Acronym: PIONEER 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4234; 2015-005326-19 (EudraCT Number); U1111-1176-9230 (Other: WHO)
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral administration once daily.
  Arms: Semaglutide
Drug: placebo — Oral administration once daily.
  Arms: Placebo

SUMMARY:
This trial is conducted globally. The aim of this trial is to investigate efficacy and safety of oral semaglutide versus placebo in subjects with type 2 diabetes and moderate renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus for at least 90 days prior to day of screening
* HbA1c (glycosylated haemoglobin) of 7.0-9.5% (53-80 mmol/mol) (both inclusive)
* Moderate renal impairment defined as estimated glomerular filtration rate of 30-59 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula
* Stable daily dose(s) within 90 days prior to the day of screening of any of the following treatment regimens:
* 1-2 of the following oral anti-diabetic drugs:
* Metformin equal or above 1500 mg or maximum tolerated dose documented in the subject medical record),
* Sulfonylurea (equal or above half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record)
* Basal insulin alone (20% change in total daily dose of insulin glargine, insulin detemir, insulin degludec or NPH insulin) or
* Metformin (equal or above 1500 mg or maximum tolerated dose documented in the subject medical record) in combination with basal insulin (20% change in total daily dose of insulin glargine, insulin detemir, insulin degludec or NPH insulin)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice). For certain specific countries: Additional specific requirements apply
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroid Carcinoma
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation
* Subjects presently classified as being in New York Heart Association Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with alanine aminotransferase above 2.5 x upper normal limit
* Rapidly progressing renal disease (e.g. such as acute glomerulonephritis) as judged by the investigator or known nephrotic albuminuria (above 2200 mg/24 hours or above 2200 mg/g)
* Use of systemic immunosuppressive treatment within 90 days prior to screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days
* Known hypoglycaemic unawareness and/or recurrent severe hypoglycaemic episodes as judged by the investigator
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (107):
- United States (55):
  - Novo Nordisk Investigational Site, Tuscumbia, Alabama
  - Novo Nordisk Investigational Site, Bermuda Dunes, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Costa Mesa, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Danbury, Connecticut
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Marietta, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Avon, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Teaneck, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, New Hyde Park, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
- Denmark (7):
  - Novo Nordisk Investigational Site, Aalborg
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, København S
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Svendborg
- Finland (7):
  - Novo Nordisk Investigational Site, Ähtäri
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Turku
- Israel (6):
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Rehovot
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Poland (2):
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Zabrze
- Russia (15):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Belgorod
  - Novo Nordisk Investigational Site, Chelyabinsk
  - Novo Nordisk Investigational Site, Dzerzhinskiy
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ulyanovsk
  - Novo Nordisk Investigational Site, Volgograd
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yaroslavl
  - Novo Nordisk Investigational Site, Yoshkar-Ola
- Sweden (6):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Skövde
  - Novo Nordisk Investigational Site, Uppsala
  - Novo Nordisk Investigational Site, Vindeln
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Bexhill-on-Sea
  - Novo Nordisk Investigational Site, Doncaster
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Milton Keynes
  - Novo Nordisk Investigational Site, Rothwell
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Wellingborough

IPD SHARING:
Plan to Share IPD: Yes
According to Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Mosenzon O, Blicher TM, Rosenlund S, Eriksson JW, Heller S, Hels OH, Pratley R, Sathyapalan T, Desouza C; PIONEER 5 Investigators. Efficacy and safety of oral semaglutide in patients with type 2 diabetes and moderate renal impairment (PIONEER 5): a placebo-controlled, randomised, phase 3a trial. Lancet Diabetes Endocrinol. 2019 Jul;7(7):515-527. doi: 10.1016/S2213-8587(19)30192-5. Epub 2019 Jun 9. PMID 31189517
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Mosenzon O, Capehorn MS, De Remigis A, Rasmussen S, Weimers P, Rosenstock J. Impact of semaglutide on high-sensitivity C-reactive protein: exploratory patient-level analyses of SUSTAIN and PIONEER randomized clinical trials. Cardiovasc Diabetol. 2022 Sep 2;21(1):172. doi: 10.1186/s12933-022-01585-7. PMID 36056351
- [Derived] Pratley RE, Crowley MJ, Gislum M, Hertz CL, Jensen TB, Khunti K, Mosenzon O, Buse JB. Oral Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Glucose-Lowering Medication: PIONEER Subgroup Analyses. Diabetes Ther. 2021 Apr;12(4):1099-1116. doi: 10.1007/s13300-020-00994-9. Epub 2021 Mar 4. PMID 33660198
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 8 countries (107 sites screened/88 randomised subjects), as follows: Denmark: 7/4; Finland: 7/7; Israel: 7/6; Poland: 2/2; Russian Federation: 19/18; Sweden: 6/4; United Kingdom: 9/7; United States (US):50/40. In addition, 10 sites in the US were approved by the institutional review board, but didn't randomise any subject
Pre-assignment Details: Data presented in "participant flow" is based on the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Groups:
- Oral Semaglutide 14 mg: Participants were to take oral semaglutide tablets once daily in a dose escalation manner from week 0 to week 26: 3 mg from week 0 to week 4, 7 mg from week 4 to week 8 and 14 mg from week 8 to week 26.
- Placebo: Participants were to take oral semaglutide placebo tablets once daily from week 0 to week 26.
Period: Overall Study
Arm/Group | Oral Semaglutide 14 mg | Placebo
Started | 163 | 161
Full Analysis Set (FAS) | 163 | 161
Safety Analysis Set (SAS) | 163 | 161
Completed | 158 | 156
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 2

BASELINE CHARACTERISTICS:
Population: The FAS comprised all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide 14 mg | Placebo | Total
Number analyzed (Participants) | 163 | 161 | 324
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71 (8) | 70 (8) | 70 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 88 | 168
  Male | 83 | 73 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 14 | 21
  Not Hispanic or Latino | 156 | 147 | 303
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 9 | 13
  White | 158 | 152 | 310
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.0 (0.7) | 7.9 (0.7) | 8.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Percentage of HbA1c
  In-trial: number analyzed (Participants) | 154 | 155
  In-trial | -1.1 (1.0) | -0.2 (0.9)
  On-treatment without rescue medication: number analyzed (Participants) | 126 | 127
  On-treatment without rescue medication | -1.2 (0.9) | -0.1 (0.9)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an analysis of covariance (ANCOVA) model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -0.8, 95% CI 2-sided [-1.0 to -0.6] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata, interaction strata and region as categorical fixed effects and the baseline value as covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.0, 95% CI [-1.2 to -0.8] — Oral semaglutide 14 mg - Placebo

2. Secondary Outcome: Change in Body Weight (kg)
Description: Change from baseline (week 0) in body weight was evaluated at week 26. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
kg
  In-trial: number analyzed (Participants) | 154 | 155
  In-trial | -3.5 (3.8) | -0.9 (2.9)
  On-treatment without rescue medication: number analyzed (Participants) | 126 | 127
  On-treatment without rescue medication | -3.9 (3.6) | -0.9 (2.9)
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 26 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using an ANCOVA model with treatment, strata, and region as categorical fixed effects and baseline body weight value as covariate for each of the 1000 imputed complete data sets, and pooled by Rubin's rule to draw inference; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern Mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -2.5, 95% CI 2-sided [-3.2 to -1.8] — Oral semaglutide 14 mg - Placebo
Statistical Analysis 2: Comparison: Oral Semaglutide 14 mg vs Placebo; The analysis was based on a MMRM that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 26. The independent effects were treatment, strata, interaction strata and region as categorical fixed effects and the baseline value as covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, MMRM — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -2.7, 95% CI 2-sided [-3.5 to -1.9] — Oral semaglutide 14 mg - Placebo

3. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 151 | 151
mmol/L | -1.58 (2.96) | -0.34 (3.03)

4. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Percentage change | -3.75 (4.10) | -0.92 (3.13)

5. Secondary Outcome: Change in BMI
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
kg/m^2 | -1.2 (1.3) | -0.3 (1.0)

6. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Centimetre (cm)
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 152 | 154
Centimetre (cm) | -2.8 (4.9) | -0.7 (3.8)

7. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol), ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 89 | 35
  No | 65 | 120

8. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol), AACE Target (Yes/no)
Description: Participants who achieved HbA1c ≤6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no), was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 60 | 12
  No | 94 | 143

9. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss ≥5% of their baseline body weight (yes/no) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 55 | 15
  No | 99 | 140

10. Secondary Outcome: Participants Who Achieve Weight Loss ≥10% (Yes/no)
Description: Participants who achieved weight loss of ≥10% of their baseline body weight (yes/no) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 13 | 0
  No | 141 | 155

11. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c <7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) was evaluated at week 26. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 78 | 27
  No | 76 | 128

12. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction ≥1% and weight loss of ≥3% (yes/no) was evaluated at week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 154 | 155
Participants
  Yes | 60 | 12
  No | 94 | 143

13. Secondary Outcome: Change in Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in total cholesterol (mmol/L) at week 26 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 148 | 153
Ratio of total cholesterol | 0.97 (20.1) | 1.00 (23.0)

14. Secondary Outcome: Change in LDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in low-density lipoprotein (LDL) cholesterol (mmol/L) at week 26 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 148 | 152
Ratio of LDL cholesterol | 0.97 (32.7) | 1.00 (38.2)

15. Secondary Outcome: Change in HDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in high-density lipoprotein (HDL) cholesterol (mmol/L) at week 26 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 148 | 153
Ratio of HDL cholesterol | 1.02 (17.5) | 1.02 (15.4)

16. Secondary Outcome: Change in Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in triglycerides (mmol/L) at week 26 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 148 | 153
Ratio of triglycerides | 0.87 (37.7) | 0.95 (37.1)

17. Secondary Outcome: Change in CRP (Ratio to Baseline)
Description: Change from baseline (week 0) in C-reactive protein (CRP) (mg/L) at week 26 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of CRP
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 152 | 154
Ratio of CRP | 0.86 (135.1) | 1.00 (136.0)

18. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the period, from week 0 to week 26. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 26), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants | 12 | 21
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, interaction strata, and region as categorical fixed effects and baseline HbA1c as covariate. Withdrawal for any reason or lost to follow-up contributed to the analysis as events (initiation of additional anti-diabetic medication). Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.1834, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.34 to 1.23]

19. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the period, from week 0 to week 26. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-26
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants | 7 | 16
Statistical Analysis 1: Comparison: Oral Semaglutide 14 mg vs Placebo; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment, strata, interaction strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0610, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.17 to 1.04]

20. Secondary Outcome: Number of TEAEs
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Events | 463 | 331

21. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG-confirmed symptomatic hypoglycaemic episodes were recorded from week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Hypoglycaemic episodes with onset during the first dose of trial product until last dose of trial product were considered treatment -emergent. Severe or BG-confirmed symptomatic hypoglycaemia was defined as an episode, that is severe according to the ADA classification or BG-confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Episodes | 17 | 3

22. Secondary Outcome: Participants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes (Yes/no)
Description: Number of participants with treatment emergent severe or BG-confirmed symptomatic hypoglycaemic episodes was recorded from week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Hypoglycaemic episodes with onset during the first dose of trial product until last dose of trial product were considered treatment -emergent. Severe or BG-confirmed symptomatic hypoglycaemia was defined as an episode, that is severe according to the ADA classification or BG-confirmed by a plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-31
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants | 9 | 3

23. Secondary Outcome: Change in Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in amylase (units/litre (U/L)) at week 26 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 129 | 140
Ratio of amylase | 1.09 (22.9) | 0.99 (25.6)

24. Secondary Outcome: Change in Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (U/L) at week 26 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 129 | 140
Ratio of lipase | 1.16 (57.6) | 0.94 (52.5)

25. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at week 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 133 | 141
Beats/minute | 1 (9) | -1 (9)

26. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change from baseline (week 0) in systolic and diastolic blood pressure was evaluated at week 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 133 | 141
mmHg
  Systolic blood pressure | -8 (14) | 0 (13)
  Diastolic blood pressure | -3 (9) | 0 (8)

27. Secondary Outcome: Change in Urinary Albumin to Creatinine Ratio (Ratio to Baseline)
Description: Change from baseline (week 0) in urinary albumin to creatinine ratio (mg/mmol) at week 26 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 131 | 136
Ratio | 0.86 (119.7) | 1.19 (145.4)

28. Secondary Outcome: Change in ECG
Description: Change from baseline (week 0) in electrocardiogram (ECG) was evaluated at week 26. Change from baseline results are presented as shift in findings (normal, abnormal and not clinically significant (NCS) and abnormal and clinically significant (CS)) from week 0 to week 26. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants
  Normal (week 0) to normal (week 26): number analyzed (Participants) | 52 | 48
  Normal (week 0) to normal (week 26) | 38 | 39
  Normal (week 0) to abnormal NCS (week 26): number analyzed (Participants) | 52 | 48
  Normal (week 0) to abnormal NCS (week 26) | 13 | 9
  Normal (week 0) to abnormal CS (week 26): number analyzed (Participants) | 52 | 48
  Normal (week 0) to abnormal CS (week 26) | 1 | 0
  Abnormal (week 0) NCS to normal (week 26): number analyzed (Participants) | 97 | 103
  Abnormal (week 0) NCS to normal (week 26) | 12 | 13
  Abnormal (week 0) NCS to abnormal NCS (week 26): number analyzed (Participants) | 97 | 103
  Abnormal (week 0) NCS to abnormal NCS (week 26) | 84 | 88
  Abnormal (week 0) NCS to abnormal CS (week 26): number analyzed (Participants) | 97 | 103
  Abnormal (week 0) NCS to abnormal CS (week 26) | 1 | 2
  Abnormal (week 0) CS to normal (week 26): number analyzed (Participants) | 5 | 2
  Abnormal (week 0) CS to normal (week 26) | 0 | 0
  Abnormal (week 0) CS to abnormal NCS (week 26): number analyzed (Participants) | 5 | 2
  Abnormal (week 0) CS to abnormal NCS (week 26) | 1 | 0
  Abnormal (week 0) CS to abnormal CS (week 26): number analyzed (Participants) | 5 | 2
  Abnormal (week 0) CS to abnormal CS (week 26) | 4 | 2

29. Secondary Outcome: Change in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS and abnormal CS at baseline (week [wk] -2) and wk 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system; 2) Nervous system (central and peripheral); 3) Gastrointestinal system, incl. mouth; 4) General appearance; 5) Head (ears, eyes, nose), throat, neck; 6) Lymph node palpation; 7) Musculoskeletal system; 8) Respiratory system; 9) Skin; 10) Thyroid gland.
Time Frame: Week -2, week 26
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants
  1) Cardiovascular system (wk -2): Normal | 107 | 103
  1) Cardiovascular system (wk -2): Abnormal NCS | 50 | 55
  1) Cardiovascular system (wk -2): Abnormal CS | 6 | 3
  1) Cardiovascular system (wk 26): Normal: number analyzed (Participants) | 155 | 154
  1) Cardiovascular system (wk 26): Normal | 101 | 104
  1) Cardiovascular system (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  1) Cardiovascular system (wk 26): Abnormal NCS | 48 | 47
  1) Cardiovascular system (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  1) Cardiovascular system (wk 26): Abnormal CS | 6 | 3
  2) Nervous system (wk -2): Normal | 114 | 116
  2) Nervous system (wk -2): Abnormal NCS | 41 | 45
  2) Nervous system (wk -2): Abnormal CS | 8 | 0
  2) Nervous system (wk 26): Normal: number analyzed (Participants) | 155 | 154
  2) Nervous system (wk 26): Normal | 109 | 115
  2) Nervous system (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  2) Nervous system (wk 26): Abnormal NCS | 40 | 39
  2) Nervous system (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  2) Nervous system (wk 26): Abnormal CS | 6 | 0
  3) Gastrointestinal system (wk -2): Normal | 149 | 152
  3) Gastrointestinal system (wk -2): Abnormal NCS | 14 | 9
  3) Gastrointestinal system (wk -2): Abnormal CS | 0 | 0
  3) Gastrointestinal system (wk 26): Normal: number analyzed (Participants) | 155 | 153
  3) Gastrointestinal system (wk 26): Normal | 146 | 145
  3) Gastrointestinal system (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 153
  3) Gastrointestinal system (wk 26): Abnormal NCS | 9 | 7
  3) Gastrointestinal system (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 153
  3) Gastrointestinal system (wk 26): Abnormal CS | 0 | 1
  4) General appearance (wk -2): Normal | 133 | 138
  4) General appearance (wk -2): Abnormal NCS | 27 | 20
  4) General appearance (wk -2): Abnormal CS | 3 | 3
  4) General appearance (wk 26): Normal: number analyzed (Participants) | 155 | 154
  4) General appearance (wk 26): Normal | 139 | 137
  4) General appearance (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  4) General appearance (wk 26): Abnormal NCS | 15 | 16
  4) General appearance (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  4) General appearance (wk 26): Abnormal CS | 1 | 1
  5) Head, throat, neck (wk -2): Normal | 151 | 143
  5) Head, throat, neck (wk -2): Abnormal NCS | 10 | 15
  5) Head, throat, neck (wk -2): Abnormal CS | 2 | 3
  5) Head, throat, neck (wk 26): Normal: number analyzed (Participants) | 155 | 153
  5) Head, throat, neck (wk 26): Normal | 142 | 139
  5) Head, throat, neck (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 153
  5) Head, throat, neck (wk 26): Abnormal NCS | 10 | 11
  5) Head, throat, neck (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 153
  5) Head, throat, neck (wk 26): Abnormal CS | 3 | 3
  6) Lymph node palpation (wk -2): Normal: number analyzed (Participants) | 162 | 161
  6) Lymph node palpation (wk -2): Normal | 161 | 161
  6) Lymph node palpation (wk -2): Abnormal NCS: number analyzed (Participants) | 162 | 161
  6) Lymph node palpation (wk -2): Abnormal NCS | 1 | 0
  6) Lymph node palpation (wk -2): Abnormal CS: number analyzed (Participants) | 162 | 161
  6) Lymph node palpation (wk -2): Abnormal CS | 0 | 0
  6) Lymph node palpation (wk 26): Normal: number analyzed (Participants) | 155 | 154
  6) Lymph node palpation (wk 26): Normal | 155 | 154
  6) Lymph node palpation (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  6) Lymph node palpation (wk 26): Abnormal NCS | 0 | 0
  6) Lymph node palpation (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  6) Lymph node palpation (wk 26): Abnormal CS | 0 | 0
  7) Musculoskeletal system (wk -2): Normal | 131 | 135
  7) Musculoskeletal system (wk -2): Abnormal NCS | 27 | 24
  7) Musculoskeletal system (wk -2): Abnormal CS | 5 | 2
  7) Musculoskeletal system (wk 26): Normal: number analyzed (Participants) | 155 | 153
  7) Musculoskeletal system (wk 26): Normal | 131 | 130
  7) Musculoskeletal system (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 153
  7) Musculoskeletal system (wk 26): Abnormal NCS | 22 | 21
  7) Musculoskeletal system (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 153
  7) Musculoskeletal system (wk 26): Abnormal CS | 2 | 2
  8) Respiratory system (wk -2): Normal | 154 | 150
  8) Respiratory system (wk -2): Abnormal NCS | 9 | 8
  8) Respiratory system (wk -2): Abnormal CS | 0 | 3
  8) Respiratory system (wk 26): Normal: number analyzed (Participants) | 155 | 154
  8) Respiratory system (wk 26): Normal | 151 | 147
  8) Respiratory system (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  8) Respiratory system (wk 26): Abnormal NCS | 4 | 5
  8) Respiratory system (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  8) Respiratory system (wk 26): Abnormal CS | 0 | 2
  9) Skin (wk -2): Normal | 129 | 129
  9) Skin (wk -2): Abnormal NCS | 33 | 32
  9) Skin (wk -2): Abnormal CS | 1 | 0
  9) Skin (wk 26): Normal: number analyzed (Participants) | 155 | 154
  9) Skin (wk 26): Normal | 128 | 136
  9) Skin (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  9) Skin (wk 26): Abnormal NCS | 23 | 18
  9) Skin (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  9) Skin (wk 26): Abnormal CS | 4 | 0
  10) Thyroid gland (wk -2): Normal | 150 | 146
  10) Thyroid gland (wk -2): Abnormal NCS | 12 | 15
  10) Thyroid gland (wk -2): Abnormal CS | 1 | 0
  10) Thyroid gland (wk 26): Normal: number analyzed (Participants) | 155 | 154
  10) Thyroid gland (wk 26): Normal | 142 | 140
  10) Thyroid gland (wk 26): Abnormal NCS: number analyzed (Participants) | 155 | 154
  10) Thyroid gland (wk 26): Abnormal NCS | 12 | 14
  10) Thyroid gland (wk 26): Abnormal CS: number analyzed (Participants) | 155 | 154
  10) Thyroid gland (wk 26): Abnormal CS | 1 | 0

30. Secondary Outcome: Change in Eye Examination
Description: Participants with eye examination findings, normal, abnormal NCS and abnormal CS at baseline (week -2) and week 26 are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week -2, week 26
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants
  Left eye (week -2): Normal: number analyzed (Participants) | 163 | 159
  Left eye (week -2): Normal | 57 | 66
  Left eye (week -2): Abnormal NCS: number analyzed (Participants) | 163 | 159
  Left eye (week -2): Abnormal NCS | 98 | 93
  Left eye (week -2): Abnormal CS: number analyzed (Participants) | 163 | 159
  Left eye (week -2): Abnormal CS | 8 | 0
  Left eye (week 26): Normal: number analyzed (Participants) | 151 | 150
  Left eye (week 26): Normal | 54 | 55
  Left eye (week 26): Abnormal NCS: number analyzed (Participants) | 151 | 150
  Left eye (week 26): Abnormal NCS | 92 | 95
  Left eye (week 26): Abnormal CS: number analyzed (Participants) | 151 | 150
  Left eye (week 26): Abnormal CS | 5 | 0
  Right eye (week -2): Normal: number analyzed (Participants) | 163 | 159
  Right eye (week -2): Normal | 59 | 66
  Right eye (week -2): Abnormal NCS: number analyzed (Participants) | 163 | 159
  Right eye (week -2): Abnormal NCS | 97 | 93
  Right eye (week -2): Abnormal CS: number analyzed (Participants) | 163 | 159
  Right eye (week -2): Abnormal CS | 7 | 0
  Right eye (week 26): Normal: number analyzed (Participants) | 151 | 150
  Right eye (week 26): Normal | 52 | 55
  Right eye (week 26): Abnormal NCS: number analyzed (Participants) | 151 | 150
  Right eye (week 26): Abnormal NCS | 97 | 95
  Right eye (week 26): Abnormal CS: number analyzed (Participants) | 151 | 150
  Right eye (week 26): Abnormal CS | 2 | 0

31. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies anytime during post-baseline visits (weeks 0-31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 162
Participants | 1

32. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies anytime during post-baseline visits (weeks 0-31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 162
Participants | 0

33. Secondary Outcome: Occurrence of Anti-semaglutide Binding Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide binding antibodies cross reacting with native glucagon-like peptide-1 (GLP-1) anytime during post-baseline visits (weeks 0-31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 162
Participants | 1

34. Secondary Outcome: Occurrence of Anti-semaglutide Neutralising Antibodies Cross Reacting With Native GLP-1 (Yes/no)
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Number of participants who measured with anti-semaglutide neutralising antibodies cross reacting with native GLP-1 anytime during post-baseline visits (weeks 0-31) are presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 162
Participants | 0

35. Secondary Outcome: Anti-semaglutide Binding Antibody Levels
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. It is based on the data from participants who were measured with anti-semaglutide antibodies anytime during post-baseline visits (weeks 0-31). Results are presented as percentage of bound radioactivity-labelled semaglutide /total added radioactivity-labelled semaglutide (%B/T). Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-31
Population: Overall number of participants analysed = participants who were found positive for anti-semaglutide antibodies. As only one subject was analyzed, standard deviation could not be calculated.
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 1
%B/T
  Week 4 | 3.1 (NA) — As only one subject was analyzed, standard deviation could not be calculated.
  Week 31 | 2.2 (NA) — As only one subject was analyzed, standard deviation could not be calculated.

36. Secondary Outcome: Semaglutide Plasma Concentrations for Population PK Analyses
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Semaglutide plasma concentrations were measured at weeks 4, 8, 14 and 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per litre (nmol/L)
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 163
Nanomoles per litre (nmol/L)
  Week 4: number analyzed (Participants) | 158
  Week 4 | 1.8 (113.5)
  Week 8: number analyzed (Participants) | 155
  Week 8 | 5.2 (143.4)
  Week 14: number analyzed (Participants) | 140
  Week 14 | 9.4 (206.6)
  Week 26: number analyzed (Participants) | 130
  Week 26 | 6.9 (251.3)

37. Secondary Outcome: SNAC Plasma Concentrations
Description: This outcome measure is only applicable for the oral semaglutide 14 mg treatment arm. Sodium N-[8-(2-hydroxybenzoyl) amino]caprylate (SNAC) plasma concentrations were measured after 25 and 40 minutes post-dose at weeks 4, 14 and 26. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Weeks 0-26
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Oral Semaglutide 14 mg
Number analyzed (Participants) | 163
Nanograms per milliliter (ng/mL)
  Week 4: 25 minutes post-dose: number analyzed (Participants) | 159
  Week 4: 25 minutes post-dose | 578 (347.4)
  Week 4: 40 minutes post-dose: number analyzed (Participants) | 159
  Week 4: 40 minutes post-dose | 364 (308.5)
  Week 14: 25 minutes post-dose: number analyzed (Participants) | 136
  Week 14: 25 minutes post-dose | 418 (389.7)
  Week 14: 40 minutes post-dose: number analyzed (Participants) | 137
  Week 14: 40 minutes post-dose | 330 (349.2)
  Week 26: 25 minutes post-dose: number analyzed (Participants) | 131
  Week 26: 25 minutes post-dose | 435 (688.0)
  Week 26: 40 minutes post-dose: number analyzed (Participants) | 131
  Week 26: 40 minutes post-dose | 288 (596.1)

38. Secondary Outcome: Change in Short Form Health Survey Version 2.0 (SF-36v2™, Acute Version) Health Survey: Scores From the 8 Domains and Summaries of the Physical Component Score (PCS) and the Mental Component Score (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at week 26. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Score
  1) Physical functioning: number analyzed (Participants) | 153 | 155
  1) Physical functioning | 0.71 (7.21) | -0.41 (6.43)
  2) Role functioning: number analyzed (Participants) | 153 | 155
  2) Role functioning | 1.97 (8.43) | -0.36 (7.76)
  3) Bodily pain: number analyzed (Participants) | 152 | 155
  3) Bodily pain | 3.18 (10.14) | -0.33 (11.47)
  4) General health: number analyzed (Participants) | 153 | 155
  4) General health | 0.18 (6.01) | -0.13 (5.77)
  5) Vitality: number analyzed (Participants) | 153 | 155
  5) Vitality | 0.05 (7.53) | 0.56 (8.02)
  6) Social functioning: number analyzed (Participants) | 153 | 155
  6) Social functioning | 1.87 (7.81) | -0.06 (9.64)
  7) Role emotional: number analyzed (Participants) | 153 | 155
  7) Role emotional | 0.62 (10.83) | -1.18 (12.32)
  8) Mental health: number analyzed (Participants) | 153 | 155
  8) Mental health | 0.34 (8.72) | -0.19 (9.48)
  Physical component summary (PCS): number analyzed (Participants) | 153 | 155
  Physical component summary (PCS) | 1.78 (7.16) | -0.15 (6.10)
  Mental component summary (MCS): number analyzed (Participants) | 153 | 155
  Mental component summary (MCS) | 0.26 (8.74) | -0.32 (10.15)

39. Secondary Outcome: Change in DTSQs: Individual Items and Treatment Satisfaction Score (6 of the 8 Items Summed)
Description: Change from baseline (week 0) in Diabetes Treatment Satisfaction Questionnaire - status version (DTSQs) was evaluated at week 26. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of hyperglycaemia and hypoglycaemia, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score has a minimum of 0 and a maximum of 36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction.
Time Frame: Week 0, week 26
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 152 | 154
Score
  1) Satisfaction with treatment | 0.41 (1.56) | 0.74 (1.57)
  2) Feeling of unacceptably high blood sugars | -1.26 (2.17) | -0.30 (2.08)
  3) Feeling of unacceptably low blood sugars | 0.11 (1.84) | -0.32 (1.82)
  4) Convenience of treatment | 0.43 (1.41) | 0.42 (1.76)
  5) Flexibility of treatment | 0.37 (1.45) | 0.52 (1.45)
  6) Satisfaction with understanding of diabetes | 0.31 (1.42) | 0.60 (1.59)
  7) Recommending treatment to others | 0.71 (1.73) | 0.37 (1.61)
  8) Satisfaction to continue with present treatment | 0.58 (1.84) | 0.47 (1.87)
  Total treatment satisfaction | 2.82 (6.61) | 3.13 (7.25)

40. Secondary Outcome: Change in Urinalysis
Description: Participants with urinalysis, "leukocytes and erythrocytes" findings, negative, trace, small, moderate or large at baseline (week [wk] 0) and wk 26 are presented. Participants with urinalysis, "nitrit" findings, negative or positive at baseline (wk 0) and wk 26 are presented. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week -2, week 26
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide 14 mg | Placebo
Number analyzed (Participants) | 163 | 161
Participants
  Leucocytes (wk 0): Negative: number analyzed (Participants) | 158 | 155
  Leucocytes (wk 0): Negative | 121 | 122
  Leucocytes (wk 0): Trace: number analyzed (Participants) | 158 | 155
  Leucocytes (wk 0): Trace | 14 | 7
  Leucocytes (wk 0): Small: number analyzed (Participants) | 158 | 155
  Leucocytes (wk 0): Small | 8 | 12
  Leucocytes (wk 0): Moderate: number analyzed (Participants) | 158 | 155
  Leucocytes (wk 0): Moderate | 10 | 9
  Leucocytes (wk 0): Large: number analyzed (Participants) | 158 | 155
  Leucocytes (wk 0): Large | 5 | 5
  Leucocytes (wk 26): Negative: number analyzed (Participants) | 129 | 138
  Leucocytes (wk 26): Negative | 91 | 103
  Leucocytes (wk 26): Trace: number analyzed (Participants) | 129 | 138
  Leucocytes (wk 26): Trace | 9 | 11
  Leucocytes (wk 26): Small: number analyzed (Participants) | 129 | 138
  Leucocytes (wk 26): Small | 13 | 10
  Leucocytes (wk 26): Moderate: number analyzed (Participants) | 129 | 138
  Leucocytes (wk 26): Moderate | 10 | 10
  Leucocytes (wk 26): Large: number analyzed (Participants) | 129 | 138
  Leucocytes (wk 26): Large | 6 | 4
  Erythrocytes (wk 0): Negative: number analyzed (Participants) | 158 | 155
  Erythrocytes (wk 0): Negative | 147 | 137
  Erythrocytes (wk 0): Trace: number analyzed (Participants) | 158 | 155
  Erythrocytes (wk 0): Trace | 4 | 10
  Erythrocytes (wk 0): Small: number analyzed (Participants) | 158 | 155
  Erythrocytes (wk 0): Small | 4 | 4
  Erythrocytes (wk 0): Moderate: number analyzed (Participants) | 158 | 155
  Erythrocytes (wk 0): Moderate | 1 | 1
  Erythrocytes (wk 0): Large: number analyzed (Participants) | 158 | 155
  Erythrocytes (wk 0): Large | 2 | 3
  Erythrocytes (wk 26): Negative: number analyzed (Participants) | 129 | 138
  Erythrocytes (wk 26): Negative | 115 | 122
  Erythrocytes (wk 26): Trace: number analyzed (Participants) | 129 | 138
  Erythrocytes (wk 26): Trace | 6 | 7
  Erythrocytes (wk 26): Small: number analyzed (Participants) | 129 | 138
  Erythrocytes (wk 26): Small | 6 | 3
  Erythrocytes (wk 26): Moderate: number analyzed (Participants) | 129 | 138
  Erythrocytes (wk 26): Moderate | 2 | 4
  Erythrocytes (wk 26): Large: number analyzed (Participants) | 129 | 138
  Erythrocytes (wk 26): Large | 0 | 2
  Nitrit (wk 0): Negative: number analyzed (Participants) | 158 | 155
  Nitrit (wk 0): Negative | 149 | 146
  Nitrit (wk 0): Positive: number analyzed (Participants) | 158 | 155
  Nitrit (wk 0): Positive | 9 | 9
  Nitrit (wk 26): Negative: number analyzed (Participants) | 129 | 138
  Nitrit (wk 26): Negative | 118 | 126
  Nitrit (wk 26): Positive: number analyzed (Participants) | 129 | 138
  Nitrit (wk 26): Positive | 11 | 12

ADVERSE EVENTS:
Time Frame: Week 0 to week 31 (26 weeks treatment period + 5 weeks follow-up period). Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide 14 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/163 | 2/161
Serious Adverse Events (participants affected / at risk) | 17/163 | 17/161
Other Adverse Events (participants affected / at risk) | 75/163 | 32/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=163) | Placebo (N=161)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Injection site abscess (Infections and infestations) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide 14 mg (N=163) | Placebo (N=161)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
Constipation (Gastrointestinal disorders) | 19 (23) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (24) | 6 (16)
Dyspepsia (Gastrointestinal disorders) | 16 (20) | 2 (2)
Headache (Nervous system disorders) | 10 (13) | 8 (21)
Nausea (Gastrointestinal disorders) | 31 (38) | 12 (12)
Vomiting (Gastrointestinal disorders) | 19 (29) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02827708/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT02827708/SAP_001.pdf